CLINICAL TRIAL: NCT02372162
Title: Fingerprint Characterization of Advanced HCC to Optimize Treatment Decisions and Enable an Early Prediction of Therapy Resistance (HCC Multiscale Trial-1)
Brief Title: Fingerprint Characterization of Advanced HCC
Acronym: e:Med-HCC-1
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Michael Bitzer, Deputy Director Department of Gastroenterology, University Hospital Tuebingen
Other Study IDs: e:Med Tuebingen, Protocol #1
Record Dates: First submitted 2014-10-09; First posted 2015-02-26 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; Molecular Diagnostics; Sorafenib; Therapeutic chemoembolization; Next-generation sequencing; Sequence analysis, DNA; Sequence analysis, RNA; Metabolomics
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens that will be investigated are tumor tissue and blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A - TACE: Patients with transarterial chemoembolization (TACE) will get an "Image Fingerprint" and "Molecular Fingerprint" for tumor characterization in vivo.
  Interventions: Other: Image Fingerprint; Other: Molecular Fingerprint
- Group B - Sorafenib: Patients with Sorafenib treatment will get an "Image Fingerprint" and "Molecular Fingerprint" for tumor characterization in vivo.
  Interventions: Other: Image Fingerprint; Other: Molecular Fingerprint

INTERVENTIONS:
Other: Image Fingerprint — This is an observational study that uses in depth diagnostic procedures to characterize patients with a comprehensive Image Fingerprint that includes CT, MRI and PET diagnostics
Other: Molecular Fingerprint — This is an observational study that uses in depth diagnostic procedures to characterize patients with a Molecular Fingerprint that includes next-generation sequencing

SUMMARY:
This single center, open-label, uncontrolled, non-randomized observational study in patients with advanced HCC. The patients qualify either to a local treatment with transarterial chemoembolization (TACE) or to a systemic treatment with the multikinase inhibitor sorafenib. The aim of this feasibility study is to get a comprehensive image and molecular fingerprint of individual tumors, with the intention to govern therapy decisions. Furthermore, to improve the care of patients that get progressive disease under treatment, the investigators have to improve the investigators understanding of the development of therapy resistance, which will improve patient care at the time point of progressive disease. Therefore, the data of 20 patients in each group will be used to identify molecular and / or image patterns, that can be used to predict treatment responses and thus govern an optimized individual cancer treatment for patients with advanced HCC.

DETAILED DESCRIPTION:
A single-center, open-label, uncontrolled, non-randomized clinical trial. The two treatment groups to receive:

Group A Transarterial Chemoembolization (TACE): 20 patients that are treated with TACE will get an image and molecular fingerprint of the tumor prior to the first treatment with TACE, a second image fingerprint between week 2 - 4 after the first treatment with TACE, and a third image and molecular fingerprint at the time point of progressive disease.

Group B Sorafenib: 20 patients that are treated with Sorafenib will get an image and molecular fingerprint of the tumor prior to the first treatment, between week 2 and 3 after the start of treatment and at the time point of progressive disease.

ELIGIBILITY:
Inclusion Criteria:

All inclusion criteria must be met at the time of screening unless otherwise specified:

1. Male or female ≥ 18 years.
2. Written informed consent obtained prior to any trial specific procedure.
3. Advanced stage hepatocellular carcinoma, BCLC class B for Group A and BCLC class B or C for Group B (refer to Appendix 3 for BCLC classification).
4. Child-Pugh class A and B. Only patients with Child-Pugh index class B of not more than 7 will be included. Patients with untreatable ascites or hepatic encephalopathy > Grade 1 are excluded (see exclusion criteria; (refer to Appendix 4 for Child Pugh classification)).
5. Indication for TACE or sorafenib treatment confirmed by an interdisciplinary tumor board.
6. ECOG performance status 0, 1 or 2 (refer to Appendix 2 for definitions of ECOG grades).
7. Life expectancy of 12 weeks or more.
8. Adequate hematological parameters, as demonstrated by:

   * Hemoglobin ≥ 9.0 g/dl (SI units: 5.6 mmol/l);
   * WBC ≥ 3.0 x 109/l;
   * Absolute neutrophil count ≥1,500/mm3;
   * Platelets ≥ 75 x 109/l;
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 times upper limit of normal range (ULNR);
   * Bilirubin ≤ 3 mg/dl;
   * Serum creatinine ≤ 1.5 mg/dl (SI units: 132 µmol/l);
   * Prothrombin Time (PT) International Normalized Ratio (INR) ≤ 1,5;
   * Serum potassium, magnesium and calcium within normal range.
9. Safe contraception in females of childbearing potential during the entire study using an established treatment with hormonal contraceptives for at least 2 months prior to start of screening.
10. For females of child bearing potential (without using hormonal contraceptives for at least 2 months prior to start of screening) a double contraception method is requested during the entire study meeting the criteria for an effective method of birth control. That means at least two effective birth control methods such as condoms, diaphragms or intra-uterine devices must be used.
11. Male patients with partners of child bearing potential are requested to use barrier contraception in addition to having their partner use another method of contraception during the trial and for 3 months after the last dose. Male patients will also be advised to abstain from sexual intercourse with pregnant or lactating women, or to use condoms.
12. Able to comply with all the requirements of the protocol.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for study participation:

1. Renal failure requiring hemo- or peritoneal dialysis.
2. Known central nervous system (CNS) tumors including symptomatic brain metastasis.
3. Patients with no adequate treatment for gastrointestinal bleeding and esophagus varices within 14 days prior to study entry.
4. Child-Pugh index class B in combination with more than slight ascites or hepatic encephalopathy > Grade I (see Child-Pugh index, Appendix 4).
5. History and current cardiovascular complications, including unstable angina pectoris, uncontrolled hypertension, congestive heart failure (NYHA Class III or IV) related to primary cardiac disease, a condition requiring anti arrhythmic therapy, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the trial entry.
6. Current evidence of any severe internal, psychiatric or neurologic disease.
7. Altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies.
8. Pregnant or breastfeeding women.
9. Active alcohol and/or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18, of both genders, with advanced stage hepatocellular carcinoma, for Group A BCLC class B (intermediate stage, performance status-ECOG 0, multinodular HCC), for Group B BCLC class B or C (advanced stage, performance status-ECOG 1-2, invasive tumor pattern (vascular invasion/extra hepatic spread)).
  Number: Up to 20 patients to receive therapy with TACE (Group A) and up to 20 patients to receive Sorafenib as first-line systemic therapy (Group B).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Availability of comprehensive imaging and molecular fingerprint data of individual tumors | Each patient will be evaluated within six months, the whole study outcome will need 48 months
  The aim of this feasibility study is to get comprehensive image and molecular fingerprints of individual tumors that can be used for systems biology approaches to predict therapy outcome and govern therapeutic decisions.

SECONDARY OUTCOMES:
Determination of turnaround time for image and molecular data availability | Each patient will be evaluated within six months, the whole study outcome will need 48 months
  To set-up and optimize the workflow of data gathering and analysis for molecular and image fingerprints.
Description of correlations between image and molecular data | Each patient will be evaluated within six months, the whole study outcome will need 48 months
  Correlation of results from image and molecular fingerprints at one point of time
Description of correlations between image and molecular data | Each patient will be evaluated within six months, the whole study outcome will need 48 months
  Correlation of either image or molecular fingerprints at three different time points
Identification of molecular and image patterns of treatment failure | Each individual patient will be evaluated within six months, the whole study outcome will need 48 months
  To identify molecular and image patterns of early treatment failure.
Identification of molecular and image patterns of treatment success | Each individual patient will be evaluated within six months, the whole study outcome will need 48 months
  To identify molecular and image patterns of early treatment success
Comparison of molecular and image pattern fingerprints in patients and animal models | Evaluation within 48 months
  To compare molecular and image patterns from HCC patients with respective patterns from different animal models which might identify suitable preclinical models for different clinical tumor patterns.
Identification of early outcome prediction patterns | Evaluation within 48 months
  To determine ideal imaging methods for an early prediction of progressive disease
To provide data for a molecular diagnostic board | Each individual patient will be evaluated as soon as data sets are available within this feasibility study
  To set up a molecular diagnostic board that checks for data-based tailored treatment options
Biomarker analysis | Evaluation within 48 months
  To identify clinical relevant biomarkers from tumor tissue or blood / urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bitzer, MD, Principal Investigator — University Clinic, Eberhard Karls University, Tübingen, Germany
Locations (1):
- University Hospital, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Homepage University Tübingen, Department of Internal Medicine I — http://im1-tuebingen.de